CLINICAL TRIAL: NCT02347631
Title: A Comparison of the Effects of Alcon DAILIES TOTAL1 and a Control High Oxygen Permeable Silicone Hydrogel Daily Disposable Contact Lens, the ACUVUE TruEye, on the Biology of the Ocular Surface and Lid Margin.
Brief Title: DAILIES TOTAL1 Versus ACUVUE TruEye - Effects on the Biology of the Ocular Surface and Lid Margin
Acronym: TruEyeTotal1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Danielle Robertson, O.D., Ph.D - Clinician Scientist, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU112014-068
Record Dates: First submitted 2015-01-15; First posted 2015-01-27 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-11

CONDITIONS: Soft Contact Lenses; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Alcon DAILIES TOTAL1, and ACUVUE TruEye (Experimental): Intervention: Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Interventions: Device: Soft Contact Lens - Daily Disposable Alcon Dailies Total 1 and ACUVUE TruEye
- ACUVUE TruEye and Alcon Dailies Total 1 (Active Comparator): Intervention: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Interventions: Device: Soft Contact Lens - Acuvue TruEye and Alcon DAILIES TOTAL 1.

INTERVENTIONS:
Device: Soft Contact Lens - Daily Disposable Alcon Dailies Total 1 and ACUVUE TruEye — Soft contact lens - Daily wear disposable lens to correct myopia in subjects who are nearsighted. Comparison of Alcon Dailies Total 1 versus Acuvue TruEye when worn as daily disposables over a two month period. This is a cross-over study where both brands of lenses will be worn by each participant over the course of the trial. Participants will be randomized for the order in which the two brands of lenses will be worn. There is a washout period of one month in between each 2 month contact lens wearing period.
  In this experimental arm, Alcon Dailies Total 1 lenses will be worn first.
  Arms: Alcon DAILIES TOTAL1, and ACUVUE TruEye
Device: Soft Contact Lens - Acuvue TruEye and Alcon DAILIES TOTAL 1. — Soft contact lens - Daily wear disposable lens to correct myopia in subjects who are nearsighted. Comparison of Alcon Dailies Total 1 versus Acuvue TruEye when worn as daily disposables over a two month period. This is a cross-over study where both brands of lenses will be worn by each participant over the course of the study. Participants will be randomized for the order in which the two brands of lenses will be worn. There is a washout period of one month in between each 2 month contact lens wearing period.
  In this active comparator arm, Acuvue TruEye lenses will be worn first.
  Arms: ACUVUE TruEye and Alcon Dailies Total 1

SUMMARY:
This is a prospective, single center, randomized, bilateral crossover, dispensing clinical trial to evaluate the effects of the water gradient lens, DAILIES TOTAL1, on the biology of corneal epithelium over two months of daily wear compared to wear of a control high oxygen permeable silicone hydrogel daily disposable contact lens, the ACUVUE TruEye; and to correlate these changes with alterations in the lid wiper, tear film and cellular changes at the limbus. The total proposed duration of this study is 12 months to ensure enrollment of up to 94 established contact lens wearers, with anticipated completion of 84. Data will be collected at baseline and following 2 months of daily wear for each lens type. Based upon data from the investigators previous contact lens clinical trials, a 1 month washout period is required prior to initiating lens wear and also between lens wear periods for the two types of lenses in order to eliminate any potential residual solution or lens effects on the corneal epithelium and restore homeostasis. The study is scheduled to commence upon Institutional Review Board approval.

DETAILED DESCRIPTION:
The following Standard of Care procedures will be performed during this study:

I.Medical history and Concomitant Medication Recorded - Subjects will be interviewed about their demographics, medical and ocular History, and their allergies and medications. The study doctor or the study personnel will use paper source documents (Case Report Form) to collect and record the following data: current prescription of both contact lenses and glasses, refraction, and keratometry.

II.Comprehensive Exam

A. Snellen visual acuity testing (both eyes) This will be performed using a standard projector chart at twenty feet. All patients will be refracted to ensure that visual acuity and prescription are within the inclusion criteria.

B. Anterior ocular segment inspection by slit lamp examination

1. Blink rate is estimated per minute (both eyes)
2. Normal eyelid and eyelash position is checked for both upper and lower lids (both eyes)
3. The tear meniscus is inspected and estimated for height in millimeter and presence or absence of cells and debris including mucous threads (both eyes)
4. The bulbar conjunctiva, cornea, anterior chamber, iris, and crystalline lens are inspected for any abnormalities (both eyes)
5. Meibomian gland orifices are inspected for signs of inflammation or plugging; eyelid skin margin is inspected for inflammation and scaling (both eyes).

C. Aqueous tear production (both eyes) Following application of 1 drop of topical tetracaine, Schirmer test strips are applied to the lower fornix at the outer one-third of the lower eyelid for 3 minutes and the length of wetting recorded in mm (≥ 3.0 mm wetting/3 minutes considered within normal limits).

D. Corneal staining (both eyes) One-drop of non-preserved isotonic saline is placed upon the tip of a fluorescein test strip and applied to the lower fornix with the patient looking up; presence or absence of corneal staining with fluorescein is then noted by the screening clinician.

E. Intraocular pressure measurement One drop of tetracaine is applied and the cornea is gently applanated with the tip of the Goldmann tonometer to ensure Intraocular pressure ≤ 21 mmHg (both eyes).

F. Evaluation of upper and lower eyelids Both upper eyelids are gently everted and both upper and lower conjunctival surfaces inspected for any abnormalities.

G. Fundus examination The pupil is dilated OU (both eyes) with 1 drop each of 2.5% neosynephrine and 0.15% mydriacyl applied 1x, X2, or x3 as needed at 10 minute intervals to achieve >5 mm dilation OU. The fundus is then inspected for the appearance of the optic nerve, macula, retinal vessels and periphery and any abnormalities noted. Any abnormalities are cause for non-inclusion.

The following Experimental Procedures will be performed:

I. Informed Consent Process The research staff will review the study including the informed consent in detail and allow the subject time to make an informed decision. Following review and opportunity to ask questions, the subject will be asked to sign this consent form.

II. Tear collection (both eyes) Tear collection will be performed as the first clinical test. Three µl sample volumes tears will be collected non-invasively in vivo using microcapillary tubes from the inferior tear meniscus at the temporal canthus of both eyes. Tears will be collected with the patient seated at the slit lamp with the light on low illumination.

III. Corneal epithelial cell collection (left eye only) Corneal epithelial cells can be collected non-invasively in vivo using a custom-made ocular irrigation chamber specific for these types of studies. The corneal irrigation chamber collects corneal epithelial cells into a 15 ml test tube. The patient is seated with forehead resting against a headrest; a fixation target is placed to orient the eye to be irrigated downwards; and the irrigating tip is positioned 2 mm below the corneal apex. Irrigation involves the delivery of 9 ml of sterile saline to the central cornea for a period of 1 minute via a tubing pump.

IV. In vivo confocal microscopy (right eye) A Heidelberg confocal microscope engineered in house with remote controlled scanning capabilities will be utilized in this study. One drop of topical tetracaine will be placed in the subject's eye; the subject's head is then placed in the headrest as for regular slit lamp examination. A drop of Genteal (Alcon Laboratories) is placed upon the top of the objective lens to serve as an immersion fluid. The cornea is then applanated using the standard objective lens tip. Both confocal microscopy through focusing scans and static images of the corneal epithelial surface will be acquired in the central cornea and all four quadrants of the limbus by controlling for the patient's direction of gaze. Similar image sequences will be performed to sequentially image the upper and lower lid wiper region at the midpoint of the eyelid (corresponding to the 5 and 7 o'clock position of the limbus). For upper lid imaging, the lid will be everted prior to image acquisition. Sequential imaging will allow for subsequent montage generation of the mid-point of the upper and lower lid.

Per visit details:

Visit 1: Screening Visit - Comprehensive ocular examination (Contact Lens Clinic at UTSW) (This visit will last ~ 90 minutes)

1. Informed Consent reviewed and signed
2. Medical History and Concomitant Meds
3. Comprehensive examination
4. Back-up glasses ordered as needed
5. Lens fitting and ordering based on randomization into the following lens groups:

   Alcon DAILIES TOTAL1 Johnson and Johnson ACUVUE TruEye
6. One month washout begins

Visit 2: Baseline Visit, lens 1 dispensed (This visit will last ~ 60 minutes)

1. Brief screening exam (go over medical history, medications, and slit lamp exam)
2. Informed consent re-reviewed
3. Baseline biological indicators (outcome measures) assessed Tear collection OU (OU = both eyes) Lid wiper staining OD (OD = Right eye) Ocular irrigation (collect epithelial cells) OS (OS = Left eye) Confocal microscopy of cornea, limbus and lid margin OD
4. Lenses dispensed

Visit 3: 1 week of lens wear (+/- 3 days) (This visit will last ~ 30 minutes)

1. Contact lens check up

   1. Lens fitting
   2. Slit lamp examination without corneal staining

Visit 4: 2 month of lens wear (+/- 3 days) (This visit will last ~ 60 minutes)

1. Brief screening exam (go over medical hx, medications, and slit lamp exam)
2. Lenses and diaries collected
3. Biological indicators assessed

i. Lenses collected OU ii. Tear collection OU iii. Lid wiper staining OD iv. Ocular irrigation OS v. Confocal microscopy of cornea, limbus and lid margin OD d. Patient begins next 1 month washout period

Visit 5: Baseline visit, lens 2 dispensed (This visit will last ~ 60 minutes) a. Brief screening exam (go over medical hx, medications, and slit lamp exam) b. Baseline biological indicators assessed i. Lenses collected OU ii. Tear collection OU iii. Lid wiper staining OD iv. Ocular irrigation OS v. Confocal microscopy of cornea, limbus and lid margin OD c. Lenses dispensed - begin crossover phase

Visit 6: 1 week of lens wear (+/- 3 days) (This visit will last ~ 30 minutes)

a. Contact lens check up

1. Lens fitting
2. Slit lamp examination without corneal staining

Visit 7: 2 month of lens wear (+/- 3 days) (This visit will last ~ 60 minutes)

1. Brief screening exam (go over medical hx, medications, and slit lamp exam)
2. Lenses and diaries collected
3. Biological indicators assessed

i. Lenses collected OU ii. Tear collection OU iii. Lid wiper staining OD iv. Ocular irrigation OS v. Confocal microscopy of cornea, limbus and lid margin OD d. Study completed

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-38 years
* Any sex, race or national origin accepted as with our past studies. Minority representation will be proactively encouraged
* Sign written informed consent
* A habitual contact lens wearer and only wear lenses for daily wear use (no overnight wear)
* Myopia range: -1.00 to -6.00 with regular astigmatism (≤1 Diopter, both eyes)
* Be willing to wear spectacles for two 1-month washout periods
* Have acceptable fit with test lenses and be willing to wear lenses for the duration of the study.
* Need correction in both eyes and be correctable to within 3 letters (high contrast Snellen VA) of their current contact lens prescription at baseline in each eye with the test lenses.
* No history of allergic eye disease either seasonal or associated with previous contact lens wear.
* A routine screening complete ocular examination (COE) with ocular findings considered to be within normal limits.
* Be willing and able to follow instructions regarding the wear of the daily disposable lenses and attend the scheduled follow-up visits.
* Must be able to arrange weekday appointments between 8:00 (morning) and 12:00 (noon).

Exclusion Criteria:

* Habitual lens wearers unable to wear lenses for a minimum of 8 hours per day.
* Use of concurrent ocular medication
* Habitual toric or bifocal contact lens wearers
* Any previous history of keratorefractive surgery or recent ocular injuries or ocular surgery within the prior 3 months
* Any preexisting ocular disease
* Monocular contact lens wear
* Any systemic disease or ocular abnormality that may impact optimal contact lens wear
* Use of systemic medications including but not limited to antihistamines, corticosteroids, anticholinergics or immunomodulatory agents
* Pregnancy or lactation
* Concurrent enrollment in another clinical trial

Ages: 21 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2016-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Robertson, O.D., PhD, Principal Investigator — UTSW Medical Center
Locations (1):
- Aston Ambulatory Care Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou S, Robertson DM. Wide-Field In Vivo Confocal Microscopy of Meibomian Gland Acini and Rete Ridges in the Eyelid Margin. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):4249-4257. doi: 10.1167/iovs.18-24497. PMID 30128496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for eligibility in 2017 at the Aston Ambulatory Optometry Clinic at UT Southwestern Medical Center.
Pre-assignment Details: 118 patients were randomize for the study. This is a crossover to compare patients who wear DAILIES contact lenses first, then TruEye contact lenses, vs. patients who wear TruEye contacts first, them DAILIES contact lenses second.
Groups:
- Alcon DAILIES TOTAL1, Then ACUVUE TRUEYE Contact Lenses: Comparison of Alcon Dailies Total 1 versus Acuvue TruEye when worn as daily disposables over a two month period. This is a crossover project where both lenses will be worn by participant over the course of the study. The order of randomization will differ for each participant.
  Intervention 1: Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Washout period - 1 month
  Intervention 2: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
- ACUVUE TRUEYE, Then Alcon DAILIES TOTAL1 Contact Lenses: Comparison of Acuvue TruEye versus Alcon Dailies Total 1 contact lenses when worn as daily disposables over a two month period. This is a crossover project where both lenses will be worn by participant over the course of the study. The order of randomization will differ for each participant.
  Intervention 1: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Washout period - 1 month
  Intervention 2 : Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
Period: Washout 1 (1 Month)
Arm/Group | Alcon DAILIES TOTAL1, Then ACUVUE TRUEYE Contact Lenses | ACUVUE TRUEYE, Then Alcon DAILIES TOTAL1 Contact Lenses
Started | 61 | 57
Completed | 61 | 57
Not Completed | 0 | 0
Period: First Intervention (2 Months)
Arm/Group | Alcon DAILIES TOTAL1, Then ACUVUE TRUEYE Contact Lenses | ACUVUE TRUEYE, Then Alcon DAILIES TOTAL1 Contact Lenses
Started | 61 | 57
Completed | 54 | 51
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Moved out of area | 0 | 2
Not completed — Lost to Follow-up | 5 | 3
Period: Washout 2 (1 Month)
Arm/Group | Alcon DAILIES TOTAL1, Then ACUVUE TRUEYE Contact Lenses | ACUVUE TRUEYE, Then Alcon DAILIES TOTAL1 Contact Lenses
Started | 54 | 51
Completed | 52 | 48
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: Second Intervention (2 Months)
Arm/Group | Alcon DAILIES TOTAL1, Then ACUVUE TRUEYE Contact Lenses | ACUVUE TRUEYE, Then Alcon DAILIES TOTAL1 Contact Lenses
Started | 52 | 48
Completed | 39 | 44
Not Completed | 13 | 4
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alcon DAILIES TOTAL1, and ACUVUE TRUEYE Contact Lenses: Comparison of Alcon Dailies Total 1 versus Acuvue TruEye when worn as daily disposables over a two month period. This is a crossover project where both lenses will be worn by participant over the course of the study. The order of randomization will differ for each participant.
  Intervention 1: Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Washout period - 1 month
  Intervention 2: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
- ACUVUE TRUEYE, and Alcon DAILIES TOTAL1 Contact Lenses: Comparison of Acuvue TruEye versus Alcon Dailies Total 1 contact lenses when worn as daily disposables over a two month period. This is a crossover project where both lenses will be worn by participant over the course of the study. The order of randomization will differ for each participant.
  Intervention 1: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
  Washout period - 1 month
  Intervention 2 : Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
- Total: Total of all reporting groups
Arm/Group | Alcon DAILIES TOTAL1, and ACUVUE TRUEYE Contact Lenses | ACUVUE TRUEYE, and Alcon DAILIES TOTAL1 Contact Lenses | Total
Number analyzed (Participants) | 61 | 57 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 57 | 118
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 81
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 51 | 46 | 97
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 20 | 17 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 25 | 29 | 54
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 7 | 4 | 11
Desquamation rate [Mean (Standard Deviation); unit: cells/min] | 76.98 (21.97) | 79.26 (20.88) | 78.72 (21.32)

OUTCOME MEASURES:

1. Primary Outcome: Desquamation Rate of Wearing Alcon DAILIES, Then AcuVue TruEye Contact Lenses
Description: Group 1: Rate of desquamation of corneal epithelial cells (cells/min) will be assessed for participants wearing Alcon DAILIES contacts lenses.
  1. Initial 1 mo. washout period (baseline 1).
  2. Participant wears the Alcon DAILIES contacts for 2 months after baseline 1.
  Group 2: Rate of desquamation of corneal epithelial cells (cells/min) will be assessed for participants wearing AcuVue TRUEYE contact lenses.
  1. Second 1 mo. washout period (baseline 2).
  2. Participant wears the Acuvue TRUEYE contacts for 2 months after baseline 2.
Time Frame: Baseline + 3 months
Population: All participants completed a 1 mo. washout 1 and wore the 1st set of contact lenses (Alcon DAILIES), then completed a second 1 mo. washout, and wore a 2nd set of contact lenses (Acuvue TRUEYE).
Measure: Mean (Standard Deviation); unit: cells/min
Groups:
- Alcon DAILIES TOTAL1 Contact Lenses: A 1 month washout will precede the intervention.
  Intervention: Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
- ACUVUE TRUEYE Contact Lenses: A 1 month washout will precede the intervention.
  Intervention: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
Arm/Group | Alcon DAILIES TOTAL1 Contact Lenses | ACUVUE TRUEYE Contact Lenses
Number analyzed (Participants) | 39 | 39
cells/min | 53.86 (13.00) | 54.05 (11.91)

2. Primary Outcome: Desquamation Rate of Wearing Acuvue TruEye, Then Alcon DAILIES Contact Lenses
Description: Group 1: Rate of desquamation of corneal epithelial cells (cells/min) will be assessed for participants wearing Acuvue TRUEYE contacts lenses.
  1. Initial 1 mo. washout period (baseline 1).
  2. Participant wears the Acuvue TRUEYE contacts for 2 months after baseline 1.
  Group 2: Rate of desquamation of corneal epithelial cells (cells/min) will be assessed for participants wearing Alcon DAILIES contact lenses.
  1. Second 1 mo. washout period (baseline 2).
  2. Participant wears the Alcon DAILIES contacts for 2 months after baseline 2.
Time Frame: Baseline + 3 months
Population: All participants completed a 1 mo. washout 1 and wore the 1st set of contact lenses (Acuvue TRUEYE), then completed a second 1 mo. washout, and wore a 2nd set of contact lenses (Alcon DAILIES).
Measure: Mean (Standard Deviation); unit: cells/min.
Groups:
- ACUVUE TRUEYE Contact Lenses: A 1 month washout will precede the intervention.
  Intervention 2: Soft Contact Lens - Daily Disposable Name - Acuvue TruEye Material - Narafilcon A Water Content - 46% Oxygen Permeability - 100 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 118 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm & 9.0mm Manner of Wear - Daily Disposables Wearing Time - 2 months
- Alcon DAILIES Contact Lenses: A 1 month washout will precede the intervention.
  Intervention 1: Soft Contact Lens - Daily Disposable Name - Alcon Dailies Total 1 Material - Delefilcon A Water Content - 33% Oxygen Permeability - 140 x10-11 (cm2/sec)(mL O2/mL mmHg) Oxygen Transmissibility - 156 x10-9 (cm/sec)(mL O2/mL mmHg) Base Curve - 8.5mm Manner of Wear - Daily Disposables Wearing Time - 2 months
Arm/Group | ACUVUE TRUEYE Contact Lenses | Alcon DAILIES Contact Lenses
Number analyzed (Participants) | 44 | 44
cells/min. | 53.48 (13.10) | 54.19 (12.34)

ADVERSE EVENTS:
Time Frame: Baseline + 6 months
Arm/Group | Alcon DAILIES TOTAL1 Contact Lenses | ACUVUE TRUEYE Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/118
Other Adverse Events (participants affected / at risk) | 2/118 | 0/118
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alcon DAILIES TOTAL1 Contact Lenses (N=118) | ACUVUE TRUEYE Contact Lenses (N=118)
Corneal Ulcer (Eye disorders) | 1 (1) | 0 (0)
Bacterial Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02347631/Prot_SAP_000.pdf